CLINICAL TRIAL: NCT06463197
Title: Self-acupressure for Insomnia in Perimenopausal Women: A Pilot Randomized Controlled Trial
Brief Title: Self-acupressure for Insomnia in Perimenopausal Women
Acronym: SAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, YEUNG Wing Fai, Associate professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAP
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Insomnia; Perimenopausal Women
Keywords: perimenopausal women; insomnia; sleep disorders
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers who will collect data from participants will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-acupressure group (Experimental): Subjects will attend two weekly 120-minute of self-administered acupressure training according to the group allocation in a classroom at the School Nursing, the Hong Kong Polytechnic University. The subjects will be trained to perform self-administered acupressure by an acupuncturist. To enhance interaction and ensure the quality of teaching, each class will be conducted in a small group of 5 to 7 subjects. Participants in this group will learn the self-acupressure technique and passed fidelity check. The treatment protocol included 6 acupoints, namely, Baihui (GV20) and bilateral Fenchi (GB20), Neiguan (PC6), Shenmen (HT7), Shenxu (BL23) and Yongquan (KI1) (Table 1). Subjects were given an acupressure log to record their practice at home, and they were phoned twice a week to remind their practice during the 4-week treatment period.
  Interventions: Behavioral: Self-Administered Acupressure Group
- Sleep Hygiene Education group (Active Comparator): The participants in this group will receive education on sleep hygiene. The treatment duration, frequency, and telephone follow-up schedule for the SHE group will be the same as the self-administered acupressure group (2 sessions, 2 hours each). Sleep hygiene education is often used as a comparison group in randomized controlled trials of self-help and psychological interventions for insomnia. The SHE group will provide subjects with the same amount of contact hours with the healthcare professional (instructor) in order to control the non-specific effects of practitioner-patient interaction in the self-administered acupressure group.
  Interventions: Behavioral: Sleep Hygiene Education group

INTERVENTIONS:
Behavioral: Self-Administered Acupressure Group — Subjects will attend two weekly 120-minute of self-administered acupressure training according to the group allocation in a classroom at the School Nursing, the Hong Kong Polytechnic University. The subjects will be trained to perform self-administered acupressure by an acupuncturist. To enhance interaction and ensure the quality of teaching, each class will be conducted in a small group of 5 to 7 subjects. Participants in this group will learn the self-acupressure technique and passed fidelity check. The treatment protocol included 6 acupoints, namely, Baihui (GV20) and bilateral Fenchi (GB20), Neiguan (PC6), Shenmen (HT7), Shenxu (BL23) and Yongquan (KI1) (Table 1). Subjects were given an acupressure log to record their practice at home, and they were phoned twice a week to remind their practice during the 4-week treatment period.
  Other Names: SAPG
  Arms: Self-acupressure group
Behavioral: Sleep Hygiene Education group — The participants in this group will receive education on sleep hygiene. The treatment duration, frequency, and telephone follow-up schedule for the SHE group will be the same as the self-administered acupressure group (2 sessions, 2 hours each). Sleep hygiene education is often used as a comparison group in randomized controlled trials of self-help and psychological interventions for insomnia. The SHE group will provide subjects with the same amount of contact hours with the healthcare professional (instructor) in order to control the non-specific effects of practitioner-patient interaction in the self-administered acupressure group.
  Other Names: SHEG
  Arms: Sleep Hygiene Education group

SUMMARY:
Insomnia is a common complaint in peri-menopausal women. Acupressure might be a potential way to treat insomnia. Although acupressure can be self-administered, it is uncertain that whether the effects of self-administered acupressure are comparable to that of the practitioner-administered acupressure, due to the variability in patients' capability of mastering the acupressure technique and self-compliance. Previous studies seemingly suggested that self-administered acupressure may improve sleep quality, their conclusion on the efficacy of self-administered acupressure for insomnia was limited due to the lack of standardized subjective and objective sleep assessments and unclear diagnostic method of insomnia. To fill out this research gap, the proposed study will explore the effectiveness of self-acupressure for improving sleep in perimenopasual women using an RCT approach.

DETAILED DESCRIPTION:
Insomnia is a common complaint in peri-menopausal women, with approximately one-third to half of the women aged 40-55 years suffering from insomnia. A recent clinical study indicated that the microbial composition in insomnia patients was different from healthy controls, and the immune factors and metabolic pathways could mediate the relationship between gut microbes and insomnia. However, such linkage needs more studies to verify.

Acupressure is a treatment modality in traditional Chinese medicine (TCM), in which the practitioner stimulates patient's acupoints using fingers, hands, or elbows according to TCM meridian theory.

Instead of practitioner-administered, the patients can be trained and perform acupressure on themselves. Such self-administered acupressure is less time-intensive and flexible to perform. Once the patient has learned the technique, self-administered acupressure does not cost anything, hence constitutes the lowest financial burden.

Although acupressure can be self-administered, it is uncertain that whether the effects of self-administered acupressure are comparable to that of the practitioner-administered acupressure, due to the variability in patients' capability of mastering the acupressure technique and self-compliance. Previous studies seemingly suggested that self-administered acupressure may improve sleep quality, their conclusion on the efficacy of self-administered acupressure for insomnia was limited due to the lack of standardized subjective and objective sleep assessments and unclear diagnostic method of insomnia. To fill out this research gap, the proposed study will explore the effectiveness of self-acupressure for improving sleep in perimenopasual women using an RCT approach.

ELIGIBILITY:
The inclusion criteria were as follows: (i) Chinese Hong Kong residents who were able to read Chinese; (ii) age 35 to 64 years; (iii) peri-menopausal women, defined as menstrual cycle irregularity (a change of 7 days or more in the menstrual cycle) or amenorrhea for no longer than 60 consecutive days, according to the recommendations from the Stages of Reproductive Aging Workshop; and (iv) with a current clinical DSM-5 diagnosis of insomnia disorder according to the Brief Insomnia Questionnaire. The criteria included having difficulties falling asleep, staying asleep, or early morning awakening with clinically significant consequences for daily life for at least 3 months. (v) An Insomnia Severity Index total score of at least 10 indicated that insomnia was present at the clinical level and (vi) Able to understand Chinese and Cantonese or Mandarin; (vii) willing to give informed consent and comply with the trial protocol.

For (iv) and (v), both the Brief Insomnia Questionnaire and Insomnia Severity Index were included as inclusion criteria. This is because the two scales have different purposes. Specifically, Brief Insomnia Questionnaire is used to confirm the participants fulfil the diagnostic criteria of DSM-5 insomnia disorder, while the Insomnia Severity Index is used to assess the severity of the insomnia symptoms and related daytime impairments.

The exclusion criteria are: (i) pregnancy; (ii) at significant suicide risk according to the rating by the Hamilton Depression Rating Scale item on suicide (score ≥3); (iii) no comorbid sleep disorders primarily requiring other treatments, such as sleep apnea or narcolepsy; (iv) change in the dose of their psychotropic drugs within 12 weeks prior to baseline, which would possibly indicate instability in their psychiatric condition; and (v) taking any antibiotics in 3 months before the baseline or any food containing probiotics, such as yogurt, in 7 days before the baseline.

Ages: 35 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — peri-menopausal women, defined as menstrual cycle irregularity (a change of 7 days or more in the menstrual cycle) or amenorrhea for no longer than 60 consecutive days, according to the recommendations from the Stages of Reproductive Aging Workshop
Enrollment: 40 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | Baseline
  The Insomnia Severity Index has 7 items that measured the severity of insomnia complaints and related daytime impairments. The total score ranges between 0 and 28, with the higher scores indicating more severe insomnia.
Insomnia Severity Index | Week 2
  The Insomnia Severity Index has 7 items that measured the severity of insomnia complaints and related daytime impairments. The total score ranges between 0 and 28, with the higher scores indicating more severe insomnia.
Insomnia Severity Index | Week 4
  The Insomnia Severity Index has 7 items that measured the severity of insomnia complaints and related daytime impairments. The total score ranges between 0 and 28, with the higher scores indicating more severe insomnia.

SECONDARY OUTCOMES:
A 7-day sleep diary | Measued one-week before the assessment time point.
  the subjects will be asked to record their daily sleeping-waking schedule using a standard sleep diary for 7 days, and Sleep parameters, such as sleep onset latency (SOL), wake after sleep onset (WASO), sleep efficiency (SE), and sleep duration (TST) will be measured.
Hospital Anxiety and Depression Scale | Baseline
  The Hospital Anxiety and Depression Scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Hospital Anxiety and Depression Scale | Week 2
  The Hospital Anxiety and Depression Scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Hospital Anxiety and Depression Scale | Week 4
  The Hospital Anxiety and Depression Scale is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3). It is designed to measure anxiety and depression (7 items for each subscale). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21).
Microbiota | Baseline
  16s rRNA sequencing of gut microbiota of the current study will be performed. The stool samples will be collected using commercially available kits. The kit contains a 5 ml buffer tube. The stool sample should be soaked in the buffer, therefore about 2-3 g stool will be collected. The kits will rapidly homogenize and stabilize the samples at the point-of-collection and transport and store stabilized DNA at ambient temperature for at least one month-no cold chain required.
Microbiota | Week 2
  16s rRNA sequencing of gut microbiota of the current study will be performed. The stool samples will be collected using commercially available kits. The kit contains a 5 ml buffer tube. The stool sample should be soaked in the buffer, therefore about 2-3 g stool will be collected. The kits will rapidly homogenize and stabilize the samples at the point-of-collection and transport and store stabilized DNA at ambient temperature for at least one month-no cold chain required.
Microbiota | Week 4
  16s rRNA sequencing of gut microbiota of the current study will be performed. The stool samples will be collected using commercially available kits. The kit contains a 5 ml buffer tube. The stool sample should be soaked in the buffer, therefore about 2-3 g stool will be collected. The kits will rapidly homogenize and stabilize the samples at the point-of-collection and transport and store stabilized DNA at ambient temperature for at least one month-no cold chain required.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, the Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No